CLINICAL TRIAL: NCT05017207
Title: Clinically Relevant Postoperative Pancreatic Fistula After Pancreaticoduodenectomy for Periampullary Cancer and Risk Factors: A Prospective Multicenter Study
Brief Title: Clinically Relevant Pancreatic Fistula After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Vo Truong Quoc (Other)
Responsible Party: Sponsor-Investigator, Vo Truong Quoc, Doctor, Lecturer, Surgeon, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: Trquoc
Record Dates: First submitted 2021-08-06; First posted 2021-08-23 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Fistula
Keywords: Risk factor
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with periampullary cancer and pancreaticoduodenectomy: Only one group of patient with periampullary cancer
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Pancreaticoduodenectomy with one of 2 types of pancreaticojejunal anastomosis: Blumgart and conventional duct-to-mucosa

SUMMARY:
Patients who are diagnosed with periampullary cancer will be performed pancreaticoduodenectomy with 3 types of pancreatic-jejunal anastomosis reconstructions. The investigator will analysis the complication of pancreatic fistula about: the clinical symptoms, laboratory test changing, intra-operative morphology, the risk factors

DETAILED DESCRIPTION:
This study will conduct at two centers at the same time: University of Medicine and Pharmacy Center and Cho Ray Hospital. The patients will be consulted to participate to this research from September, 2021 to April, 2023.

Plan for conducting study:

* The investigator consults and gets consensus form of the patient with periampullary cancer.
* The patient will be prepared for pancreaticoduodenectomy: pre-operative laboratory test, pre-operative biliary drainage, anesthetic checking.
* The investigator collected intr-operative data, include type of pancreatic-duodenal reconstruction, type of pancreatic duct's drainage, quantity of blood loss and blood transfusion.
* The investor follows post-operative period.
* If there are pancreatic fistula appear, the investigator will collect the clinical signs, laboratory test changing, re-operative morphology.
* The investigator analysis the risk factors of pancreatic fistula.

Data analysis:

* To determine the incidence of pancreatic fistula, the morphology of pancreatic fistula, descriptive statistics will be used.
* To determine the risk factors of pancreatic fistula, logistic regression will be used.

Sample size:

* The investigator plans to collect 145 patients in the research period.

Plan for missing data:

* Any case that miss information will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with periampullary cancer and can be performed pancreaticoduodenectomy.
* Pancreaticoduodenectomy with one of three types of pancreatic - duodenal anastomosis reconstructions.

Exclusion Criteria:

* The patient does not consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Periampullary cancer with postoperative pathology is adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pancreatic fistula | 30 days of post-operative period
  The investigator will describe the day that appears pancreatic fistula, the clinical symptoms, intra-operative morphology if being indicated to re-operate. The measurement tool to diagnose pancreatic fistula is fluid amylase on the POD3 (fluid amylse is 3 times compared to serum's amylase)
Risk factors relate to pancreatic fistula | 30 days of post-operative period
  The investigator will analyse some of the risk factors that relate to pancreatic fistula, including pre-operative factors (BMI, albumin, bilirubin, biliary drainage), intra-operative elements (pancreatic duct 's diameter, pancreatic textile, blood transfusion, portal vein reconstruction), and post-operative factors (abdominal drainage's volume, fluid amylase, abdominal abscess..). The investigator will use the multivariable regression model to determine the risk factors (p-value<0.05)

SECONDARY OUTCOMES:
Short-term result in treatment of post-operative pancreatic fistula | 30 days of post-operatvive period
  The investigator will describe the result of pancreatic fistula treatment: intra-operative morphology, re-operative success ratio, morbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Truong Quoc Vo, Principal Investigator — University of Medicine and Pharmacy at HoChiMinh City
Locations (1):
- University Medical Center of HCMC, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
The IDP will be saved as excel and spss file

REFERENCES:
- [Background] Kawaida H, Kono H, Hosomura N, Amemiya H, Itakura J, Fujii H, Ichikawa D. Surgical techniques and postoperative management to prevent postoperative pancreatic fistula after pancreatic surgery. World J Gastroenterol. 2019 Jul 28;25(28):3722-3737. doi: 10.3748/wjg.v25.i28.3722. PMID 31391768
- See also: Surgical techniques and postoperative management to prevent postoperative pancreatic fistula after pancreatic surgery — http://pubmed.ncbi.nlm.nih.gov/31391768/